CLINICAL TRIAL: NCT02141230
Title: Evaluation of the Characteristics of Alli® Purchasers in the European Union Following the Revision to the Alli® Pack Information.
Brief Title: Risk Management Plan (RMP) Survey for Purchasers of Alli® (60 mg Orlistat) in the European Union.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Hamell (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 202157; RH01159 (Other: GSK)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alli® 60 mg (Experimental): Participants purchasing Alli®
  Interventions: Drug: Alli® 60 mg

INTERVENTIONS:
Drug: Alli® 60 mg — Participants purchasing Alli®

SUMMARY:
Following results from the first survey that forms part of the EU RMP for Alli® (RMP survey 1; WEUSRTP3350), several amendments to the information included on the pack carton for Alli® (orlistat 60 mg) were recommended. The main finding from RMP survey 1 was that a large proportion of Alli® users had a body mass index (BMI) less than (<)28 kg/m2 . (Note: the European indication for Alli® is adults 18 years and older with a BMI<28 kg/m2.) The proportion of respondents overall who reported possible contraindications to Alli® use was relatively low. The following changes to the pack labeling were agreed and have been implemented: : (1) a statement, highlighting the product is only for those with a BMI of 28 or above was added to the front of the pack; (2) wording of the BMI statement on the back of the pack was strengthened; (3) contraindications were highlighted in bold text; (4) the statement that Alli® is not for use by those under 18 years of age was modified for clarity. In addition, a pharmacy reminder card was made available to retail pharmacists to improve awareness of the prescribing information for Alli®. The survey will assess whether compliance with the authorized indication and contraindications among purchasers of Alli® has been improved after one year of marketing the revised pack labeling.

ELIGIBILITY:
Inclusion Criteria:

* Any individual who purchases Alli from a pharmacy for their own personal use and provides consent.

Exclusion Criteria:

* No exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
To estimate the proportion of Alli® purchasers with a BMI <28 kg/m2. | More than one year following introduction of updated labeling.
  BMI will be calculated from self-reported weight and height measures.
To estimate the proportion of Alli® purchasers aged <18 years. | More than one year following introduction of updated labeling.
  The survey will collect the demographic details including age.

SECONDARY OUTCOMES:
To estimate the proportion of Alli® purchasers with contraindications to use (ciclosporin use, chronic malabsorption syndrome, cholestasis, pregnancy, breastfeeding, warfarin use). | More than one year following introduction of updated labeling.
  The survey will collect information on the history of contraindicated medical conditions (chronic malabsorption syndrome, cholestasis, pregnancy, breast-feeding) and use of contraindicated medications taken (ciclosporin, warfarin).
To characterise the demographic characteristics of Alli® purchasers in the EU and their patterns of previous use of over-the-counter (OTC) orlistat (defined as Alli® capsules or a generic equivalent, or alli chewable tablets). | More than one year following introduction of updated labeling.
  Demographics characteristics of the customers who have bought Alli® (capsules or chewable tablets) for their own use and the information of their previous experience with Alli® will be recorded.
To estimate the proportions of Alli® purchasers who have previously used OTC orlistat and who have a history of kidney disease or who are taking levothyroxine. | More than one year following introduction of updated labeling.
  History of kidney disease, or use of medication for hypothyroidism will be recorded in the survey for the customers who have previously used OTC orlistat.
For Alli® purchasers who have previously used OTC orlistat, descriptive data on the daily dose taken (number of capsules [or tablets]) will be collected. | More than one year following introduction of updated labeling.
  The survey will include the information on the the number of capsules (or tablets) taken per day for the customers who have previously used OTC orlistat.
To provide a descriptive comparison between the results of this survey and the previous surveys. | More than one year following introduction of updated labeling.
  Based on the information collected in the survey, a descriptive comparison will be done between the results of this survey and the previous surveys to assess whether compliance with the authorized indication and contraindications among purchasers of Alli® has been improved.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline